CLINICAL TRIAL: NCT04973241
Title: Mandibular Dimensions as a Predictor of Age and Sex in a Sample of Upper Egypt Population
Brief Title: Mandibular Dimensions as a Predictor of Age and Sex in a Sample of Upper Egypt Population by Using Panoramic Images and Cone Beam Computed Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, EMM Kotb, Eman Mahmoud Metwally, Assiut University
Other Study IDs: OPG&CBCT for mandible measures
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Mandibular Dimensions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OPG
  Interventions: Radiation: OPG & CBCT
- CBCT
  Interventions: Radiation: OPG & CBCT

INTERVENTIONS:
Radiation: OPG & CBCT — panoramic images , cone beam computed tomography

SUMMARY:
Growth changes occur from the intrauterine life to senility, hard tissues like bones and teeth undergo changes with growth, a change in shape and/or fusion of ossification centers, the stability of these changes facilitate ease in estimation of age from hard tissue samples ( Bhalaji ,2006;Reddy,2006; Mohite et al.,2011).

Mandibles were used for the study for two simple causes: First, there appears to be a lack of standards utilizing this element and second, this bone is often recovered mostly intact (Franklin et al.,2008) The mandible is considered the most durable facial bone ;is due to the presence of a dense layer of compact bone and therefore remains well conserved than many other bones and the only movable bone of the skull available for gender identification; is due to the morphological characteristics of mandible, and radiology plays an important role in it. It is composed of two hemi mandibles united at the midline by a vertical symphysis. Each one of them is composed of a horizontal body with a posterior vertical extension termed the ramus(ndira et al.,2012 ).

Mandibular canines are found to exhibit the highest sexual dimorphism.The mean age of eruption of mandibular canines is 10.87 years, and they are the last teeth to be extracted with respect to age; so, they can be considered as the key teeth for personal identification (Khangura et al.,2011; Padmavati et al.,2011; Yuwanati et al.,2012).

Measurements of the mandibular ramus tend to show higher sexual dimorphism, and variations between the sexes are mostly more marked in the mandibular ramus than in the mandibular body (Humphrey et al.,1999).

Gonial angle is commonly used to determine the rotation of the mandible and to identify growth pattern, it is a common parameter used to describe orthodontic extractions or surgical treatments(Kitai et al.,2013).

Several studies focused on the comparison between CBCT (Cone Beam Computed Tomography) and OPG (Orthopantomograph) for visualization of bone and teeth (Dalessandri et al.,2012 ;Savoldi et al.,2015).

OPG is a very popular technique ,the most available and commonly used extra-oral radiography, its lower cost ,wide area coverage ,ease of preparation have made it an excellent choice for routine examination of many structures thus useful for research purpose does not involve the patient any additional exposure or cost(Ghosh et al.,2009 ;Sairam et al.,2016).

The CBCT imaging device can obtain undistorted three-dimensional (3D) images of good quality with a low radiation dose (Yamamoto et al.,2003).

ELIGIBILITY:
Inclusion Criteria:

- 1. Panoramic radiographs and cone beam computed tomography of patients aged15-40 years.

2. Only patients with a documented date of birth.

Exclusion Criteria:

* 1. Asymmetry in OPG and CBCT images, unreadable ,unclear ,poor quality, gross pathology and magnification.

  2. Panoramic radiographs with positioning errors which could cause distortions in the dimensions.

  3. Hereditary facial asymmetries. 4. Images of completely edentulous patients. 5. Surgical intervention, patients with orthognathic surgeries. 6. Presence of pathologies such as fractures, impacted teeth, missing teeth, cleft lip or palate, cysts, tumors, osteomyelitis,severe osteoporosis in the mandible, periodontal lesion, and congenital craniofacial abnormalities, in the lower jaw, resorption in the mandibular arch that could affect the interpretation of radiographic image, 7. History of head trauma

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: persons aged between 15 and 40 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
comparison of OPG & CBCT | Baseline
  2. Comparison of the accuracy in identification of age and sex between using digital orthopantomographs and cone beam computed tomography

IPD SHARING:
Plan to Share IPD: No